CLINICAL TRIAL: NCT05981339
Title: Acute Effect of Osteopathic Visceral Mobilization Techniques on Adductor Spasticity, Incontinence and Constipation in Multiple Sclerosis Patients
Brief Title: Acute Effect of Osteopathic Visceral Mobilization Techniques
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Gaziantep (Other)
Responsible Party: Principal Investigator, Ogr Uyesi Tuba MADEN, Assisstanf Profesor, University of Gaziantep
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022/477
Record Dates: First submitted 2023-07-31; First posted 2023-08-08 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-07

CONDITIONS: Multiple Sclerosis; Pelvic Floor Disorders; Urinary Incontinence; Visceral Mobilization; Osteopathic Manipulative Treatment
MeSH Terms: conditions — Multiple Sclerosis; Pelvic Floor Disorders; Urinary Incontinence | interventions — Breathing Exercises

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial Study and Control Group
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Sham Comparator): In the control group, diaphragmatic breathing exercises will be performed together with the physiotherapist. Osteopathic manual therapy techniques will be applied as sham. The physiotherapist will not touch the appropriate anatomical points while performing the loosening.
  Interventions: Other: breathing exercises
- Study Group (Experimental): In addition to breathing exercises, sacral release and bladder mobilization, which are osteopathic manual therapy techniques, will be applied to the patients in the study group.
  Interventions: Other: breathing exercises; Other: osteopathic manual therapy techniques

INTERVENTIONS:
Other: breathing exercises — For the diaphragmatic breathing exercise, patients are asked to perform a nasal inspiration and expiration that moves predominantly the abdomen by reducing the movement of the thorax in the semi-supine position. To give tactile stimulation, one hand of the patient is placed on the chest with the other hand on the abdominal region. Continue this exercise for three minutes.
Other: osteopathic manual therapy techniques — * Sacral release: While the patient is in the side lying position, the physiotherapist goes behind the patient, one hand is placed on the lower abdominal area, and the thenar and hypothenar areas of the other hand are placed on the basis of the sacrum. It is waited until a general relaxation is felt in the tissue under the hands (Stone, C., 2006).
  * Bladder mobilization: Two hands are placed just above the pubic region and gently pressed down first to test the surface protrusion of the uterus. During the application, the pressure of the hand is adjusted according to the tension of the tissue. Hand contact is not interrupted until the fascial tissue under the hand is relaxed (Stone, C., 2006).
  Arms: Study Group

SUMMARY:
Multiple Sclerosis (MS), caused by lesions in the white matter of the central nervous system, is an autoimmune inflammatory demyelinating chronic disease.

The disease may present with many findings from fatigue, spasticity, balance and gait disturbances to bladder-bowel dysfunction (Ferreira, A.P.S., et al., 2019). When the rehabilitation methods for incontinence were examined, pelvic floor muscle training, tibial nerve stimulation and sacral neuromodulation were frequently encountered (Rahnama'I, MS., 2020). Pelvic floor muscle training should create an effective result in MS patients, and the training should be done for a long time, such as 8-12 weeks. No study has been found examining the effects of manual therapy techniques and diaphragmatic breathing exercise in the acute phase in functional or neurogenic bladder-intestinal dysfunctions.

DETAILED DESCRIPTION:
The study was planned as a randomized controlled trial. MS patients included in the study will be divided into two groups according to inclusion and exclusion criteria. Diaphragmatic breathing exercises and sacral relaxation, bladder mobilization, which are osteopathic manual therapy techniques, will be applied to the study group. On the other hand, only diaphragmatic breathing exercises will be applied to the control group.

Individuals will be treated in a single session. The acute effect of intervention will be examined by making a total of 3 evaluations, pre-intervention, post-intervention, and 1 week after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Multiple Sclerosis
* The age of 18 years and the older
* Individuals with stable medical condition
* Having complaints of urinary dysfunction for at least 6 months,
* Mini Mental test score > 24 points
* EDDS less than 6.5 (0-6.5 points will be)
* Volunteering to participate in the study

Exclusion Criteria:

* Having cognitive problems
* Presence of pelvic organ prolapse or prostate
* Pregnancy
* Abdominal surgery history
* Presence of urinary system infection
* Continuing drug use for overactive bladder
* Having received pelvic floor muscle training
* Concomitant other neurological or kidney disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-08-07 (Estimated); Primary Completion 2023-09-15 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Spasticity Assessment | Change from MAS scale at one week
  The Modified Ashworth Scale (MAS), the most common test used in clinical and research, will be used to assess spasticity. The reliability of the scale has been proven among raters in the lower extremities. According to the resistance to passive movement, the lowest score of the manual scale is 0 and the highest score is 4. The higher the score, the higher the spasticity.
Evaluation of Pelvic Floor Muscle Activity | Change from Muscle Activity scale at one week
  easurements are performed with surface electrodes and a device similar to a biofeedback device (NeuroTrac ETS™; Verity Medical, Romsey, UK) to evaluate pelvic floor muscle activity. The biofeedback device is used to train and test the pelvic floor muscles. As the values increase, so does the muscular activity.
International Consultation on Incontinence Questionnaire Short Form ICIQ-SF | Change from ICIQ-SF at one week
  To evaluate urinary incontinence and the effect of urinary incontinence on quality of life, Avery et al. The Turkish validity and reliability of the scale developed by Çetinel et al. Made by in 2004. The scale has four dimensions, in the first dimension how often urinary incontinence is, in the second dimension the amount of urinary incontinence, in the third dimension the effects of urinary incontinence on daily life and in the fourth dimension the conditions that cause urinary incontinence are questioned. The first three dimensions are scored in the evaluation. The answers given to the fourth dimension, which is not scored, are used to determine the type of urinary incontinence based on the individual's complaints. A score between 0 and 21 is obtained from the scale. A low score indicates that urinary incontinence affects the quality of life little, while a high score indicates that it affects the quality of life very much.
Constipation Quality of Life Scale: Constipation Quality of Life Scale (CIQS) | Change from CIQS at one week
  CIQS is a self-assessment scale consisting of 28 items in total, consisting of "anxiety/anxiety" (11 items), "physical discomfort" (4 items), "psycho-social discomfort" (8 items), "satisfaction" (five items). The highest score that can be obtained from the five-point Likert scale is 140, and the lowest score is 28. It is thought that the quality of life is negatively affected as the scores obtained from the scale increase.

CONTACTS AND LOCATIONS:
Locations (1):
- Tuba Maden, Gaziantep, Turkey (Türkiye)